CLINICAL TRIAL: NCT01700868
Title: Practice Based Nutrition Intervention-2
Acronym: PBNI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PBNI-2
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Diet, Vegetarian; Diet, Fat-Restricted; Glycemic Index
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Vegan; Diet, Plant-Based

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vegan Group (Experimental): Participants in the intervention group will follow a low-fat, vegan diet for 20 weeks, and will attend nutrition classes in the form of a weekly support group.
  Interventions: Other: Vegan diet
- American Diabetes Association guidelines (Active Comparator): Participants will follow ADA diet according to ADA regulations. This group will also receive weekly nutrition classes.
  Interventions: Other: American Diabetes Association guidelines

INTERVENTIONS:
Other: Vegan diet — A diet devoid of any animal products. Low-fat, low-Glycemic Index, vegan diet.
  Other Names: Plant-based diet
  Arms: Vegan Group
Other: American Diabetes Association guidelines — Participants will follow individualized diet plans following ADA guidelines
  Other Names: ADA
  Arms: American Diabetes Association guidelines

SUMMARY:
This study aims to test hypotheses that are potentially important to diabetes management, with practical implications for reducing the medical, personal, and economic costs of the disease. Anticipated outcomes include reductions in glycosylated hemoglobin that are significantly greater than those achievable with current diet recommendations, reductions in medication use among many intervention-group participants, beneficial changes in body weight and serum lipid concentrations, and a demonstration of the acceptability of the intervention diet. Progress toward these goals could refine dietary guidance for individuals with diabetes, increase treatment expectations, and reduce the massive burden the disease currently imposes.

The study further attempts to translate a dietary intervention studied in a clinical research setting to a medical practice. This will contribute to developing a model for diabetes care that can be used widely.

DETAILED DESCRIPTION:
Specific Aim 1 tests the hypothesis that the nutrition intervention (low-fat, low-GI, vegan diet; henceforth called the 'vegan diet') improves glycemic control, body weight, plasma lipid concentrations, blood pressure, and indices of renal function in a within-group analysis.

Glycosylated hemoglobin is the primary dependent variable, as well as fasting plasma glucose and urinary albumin and creatinine concentrations. The within-group changes in these variables from baseline to week 20, one-year follow-up will be compared.

Specific Aim 2 tests the hypothesis that the vegan diet is more effective than standard nutrition care for improving glycemic control, body weight, plasma lipid concentrations, blood pressure, and indices of renal function in individuals with type 2 diabetes.

Glycosylated hemoglobin is the primary dependent variable, as well as fasting plasma glucose and urinary albumin and creatinine concentrations in both the intervention and control groups. The between-groups differences in the changes in these variables from baseline to week 20, and one-year follow-up will be compared.

Specific Aim 3 tests the hypothesis that the vegan diet is sustainable among individuals with type 2 diabetes for a 20-week period, with weekly classes, and in a follow-up period of one year with limited professional support.

This will be assessed by 3-day dietary records at weeks 0, 20 and one-year follow-up.

Specific Aim 4 tests the hypothesis that the vegan diet has an acceptability that is comparable to that of standard nutrition care among individuals with type 2 diabetes.

This hypothesis will be addressed by quantitatively assessing adherence to and acceptability of the intervention and control diets, using the 3-day dietary record, the Food Acceptability Questionnaire, and the Eating Inventory, as described below.

Specific Aim 5 tests the hypothesis that the effects of the dietary interventions on A1c and body weight are reduced in individuals with the A1 and B1 alleles of the DRD2 gene.

This will be assessed through Taq1 A1 and B1 genotype determination at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of type 2 diabetes mellitus, as defined by a fasting plasma glucose concentration ≥126 mg/dl on 2 occasions or a prior physician's diagnosis of type 2 diabetes with the use of hypoglycemic medications for at least 6 months
2. male or female
3. A1c between 6.5% and 10.5%
4. age at least 18 years
5. ability and willingness to participate in all components of the study
6. willingness to be assigned to either a low-fat, vegan diet or to standard care
7. diabetes medications unchanged for 1 month prior to volunteering for the study
8. patient of Dr. Mark Sklar

Exclusion Criteria:

1. body mass index >45 kg/m2
2. alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
3. use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
4. pregnancy
5. history of severe mental illness (with current unstable status)
6. likely to be disruptive in group sessions (as determined by research staff)
7. Signs/symptoms of acute uncontrolled diabetes (including but not limited to polyuria, polydipsia, blurred vision, uncontrolled weight loss)
8. unstable medical status
9. already following a low-fat, vegetarian diet
10. an inordinate fear of blood draws
11. inability to maintain current medication regimen
12. lack of English fluency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1C (diabetes management) | 20 weeks

SECONDARY OUTCOMES:
Body Weight | 20 Weeks
Blood Pressure | 20 Weeks
Glucose | 20 Weeks
Comprehensive Metabolic Panel | 20 Weeks & one-year follow up
Serum cholesterol and triacylglycerol concentrations | 20 Weeks
Urinary albumin and creatinine | 20 Weeks
Genotyping for Taq1 A and Taq1 B polymorphisms, and APOE (Apolipoprotein E) | 20 Weeks
Waist and hip circumference | 20 Weeks
Dietary Acceptability | 20 Weeks
3-day dietary records | 20 Weeks
International Physical Activity Questionnaire | 20 Weeks
Food Acceptability Questionnaire | 20 Weeks
Eating Inventory | 20 Weeks
CESD-R (Center for Epidemiologic Studies Depression Scale: Review and revision) | 20 Weeks
Beck Depression Inventory II (BDI-II) | 20 Weeks
Height | 20 Weeks
24-Hour Multi-Pass Dietary Recalls | 20 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Esselstyn CB Jr. Updating a 12-year experience with arrest and reversal therapy for coronary heart disease (an overdue requiem for palliative cardiology). Am J Cardiol. 1999 Aug 1;84(3):339-41, A8. doi: 10.1016/s0002-9149(99)00290-8. PMID 10496449
- [Background] Nicholson AS, Sklar M, Barnard ND, Gore S, Sullivan R, Browning S. Toward improved management of NIDDM: A randomized, controlled, pilot intervention using a lowfat, vegetarian diet. Prev Med. 1999 Aug;29(2):87-91. doi: 10.1006/pmed.1999.0529. PMID 10446033